CLINICAL TRIAL: NCT01864525
Title: Effects of Octanoic Acid for Treatment of Essential Voice Tremor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Soren Lowell, Assistant Professor, Communication Sciences & Disorders, Syracuse University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 370955-3; 1R03DC012429-01A1 (NIH)
Record Dates: First submitted 2013-05-21; First posted 2013-05-29 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Essential Voice Tremor; Vocal Tremor; Voice Tremor; Essential Tremor of Voice
Keywords: voice; tremor; essential tremor; essential voice tremor; voice treatment; octanoic acid; octanol; voice disorder; dysphonia
MeSH Terms: conditions — Tremor; Essential Tremor; Voice Disorders; Dysphonia | interventions — octanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inactive capsule (Placebo Comparator): Participants will receive a pill/capsule with an inactive ingredient during the placebo arm of this study.
  Interventions: Drug: Inactive capsule
- Octanoic acid (Experimental): Participants will receive a pill/capsule with octanoic acid (amount determined by the participant's weight) during the experimental arm of this study.
  Interventions: Drug: Octanoic acid

INTERVENTIONS:
Drug: Octanoic acid
  Other Names: Caprylic acid
  Arms: Octanoic acid
Drug: Inactive capsule
  Other Names: Placebo
  Arms: Inactive capsule

SUMMARY:
Essential voice tremor is a neurological condition that produces a regular, shaking quality in the voice. One form of drug treatment that produces some improvement in tremor of the hands is octanoic acid, which is a food additive that is similar to alcohol. Research suggests that octanoic acid may reduce tremor in the hands/arms with few side effects and no intoxication effects. This study will determine whether octanoic acid may be useful for reducing tremor when it affects the voice. Researchers are hypothesizing that octanoic acid will reduce the effects of tremor on the voice.

DETAILED DESCRIPTION:
Background:

* Essential tremor of the voice produces regular shaking and hoarseness in the voice, making it difficult speech difficult to understand
* Several previous studies have found that octanoic acid and octanol, which are related to alcohol, can improve tremor in some people without producing many side effects and without producing intoxication
* Researchers are interested in determining whether octanoic acid can improve tremor that affects the voice

Objectives:

* To determine the effects of octanoic voice using voice recordings and listener ratings of voice
* To determine the effects of octanoic acid on level of voice disability experienced by people with essential voice tremor

ELIGIBILITY:
Inclusion Criteria:

* Participants have a diagnosis of essential voice tremor and show signs of tremor during the endoscopy examination (when pictures of the voice box are obtained)during screening appointment
* Participants show measurable voice tremor from recordings of the voice during screening appointment

Exclusion Criteria:

* Participants have a diagnosis or show signs of Parkinson's Disease or another non-essential tremor movement disorder
* Participants have a diagnosis or show signs of spasmodic dysphonia (a different neurological voice disorder)
* Participants have a diagnosis of a severe, non-stable medical condition, such as kidney or liver failure, severe heart disease, severe lung disease, severe metabolic disease, uncontrolled hyperthyroidism, or other life-threatening disease such as active cancer
* Participants have a diagnosis of diabetes mellitus
* Participants are unable to suspend/stop a medication that they are currently taking for tremor or voice disorder for 12 weeks to complete this study
* Participants have a dependence on alcohol or allergy to alcohol
* Participants are pregnant or lactating
* Participants have an allergy to soy
* Participants have Irritable Bowel Syndrome

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12-22 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soren Y Lowell, PhD, Principal Investigator — Syracuse University
Locations (1):
- Syracuse University & Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haubenberger D, McCrossin G, Lungu C, Considine E, Toro C, Nahab FB, Auh S, Buchwald P, Grimes GJ, Starling J, Potti G, Scheider L, Kalowitz D, Bowen D, Carnie A, Hallett M. Octanoic acid in alcohol-responsive essential tremor: a randomized controlled study. Neurology. 2013 Mar 5;80(10):933-40. doi: 10.1212/WNL.0b013e3182840c4f. Epub 2013 Feb 13. PMID 23408867
- [Result] Nahab FB, Wittevrongel L, Ippolito D, Toro C, Grimes GJ, Starling J, Potti G, Haubenberger D, Bowen D, Buchwald P, Dong C, Kalowitz D, Hallett M. An open-label, single-dose, crossover study of the pharmacokinetics and metabolism of two oral formulations of 1-octanol in patients with essential tremor. Neurotherapeutics. 2011 Oct;8(4):753-62. doi: 10.1007/s13311-011-0045-1. PMID 21594724
- [Result] Nahab FB, Handforth A, Brown T, Shin C, Quesada A, Dong C, Haubenberger D, Hallett M. Octanoic acid suppresses harmaline-induced tremor in mouse model of essential tremor. Neurotherapeutics. 2012 Jul;9(3):635-8. doi: 10.1007/s13311-012-0121-1. PMID 22454323
- [Result] Shill HA, Bushara KO, Mari Z, Reich M, Hallett M. Open-label dose-escalation study of oral 1-octanol in patients with essential tremor. Neurology. 2004 Jun 22;62(12):2320-2. doi: 10.1212/wnl.62.12.2320. PMID 15210907
- [Result] Bushara KO, Goldstein SR, Grimes GJ Jr, Burstein AH, Hallett M. Pilot trial of 1-octanol in essential tremor. Neurology. 2004 Jan 13;62(1):122-4. doi: 10.1212/01.wnl.0000101722.95137.19. PMID 14718713

RESULTS

PARTICIPANT FLOW:
Groups:
- Inactive Capsule First: Participants who were randomized to receive a capsule with an inactive ingredient (placebo) during the first 3 weeks of the study (placebo arm of crossover design study), and then received octanoic acid in the last 3 weeks of the study.
  Placebo
- Octanoic Acid First: Participants who were randomized to receive a capsule with octanoic acid (amount determined by the participant's weight) during the first 3 weeks of the study (experimental arm of crossover design study), and then received the placebo in the last 3 weeks of the study.
  Octanoic acid
Period: Overall Study
Arm/Group | Inactive Capsule First | Octanoic Acid First
Started | 10 | 7
Completed | 9 | 7
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inactive Capsule First | Octanoic Acid First | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.90 (7.20) | 70.43 (11.70) | 69.53 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 7 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 7 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of Acoustic Amplitude Tremor and Magnitude of Acoustic Frequency Tremor
Description: Voice recordings were used to measure the degree of tremor in the voice. Mean post-test values for each acoustic measure were compared after the octanoic acid and placebo conditions, with and without consideration of baseline values. Mean values represent the average of two testing days. Degree of amplitude tremor shows the extent of amplitude variation as a percent of the mean signal amplitude, with lower numbers indicating less amplitude tremor. Baseline values for magnitude of amplitude tremor across all participants and conditions ranged from 4.06 to 27.09, and post-test values ranged from 1.94 to 26.02. Degree of frequency tremor shows the extent of fundamental frequency variation as a percent of the mean signal frequency, with lower numbers indicating less frequency tremor. Baseline values for magnitude of frequency tremor across all participants and conditions ranged from 1.21 to 15.31, and post-test values ranged from 0.60 to 13.86.
Time Frame: Measured at baseline visits (1 & 2) and after 3 weeks of placebo or octanoic acid on post-test visits (1 & 2)
Measure: Mean (Standard Deviation); unit: percentage of voice signal with tremor
Groups:
- Placebo: Participants who received a capsule with an inactive ingredient (placebo) during either the first or last 3 weeks of the study.
  Placebo
- Octanoic Acid: Participants who received a capsule with octanoic acid (amount determined by the participant's weight) during either the first or last 3 weeks of the study.
  Octanoic acid
Arm/Group | Placebo | Octanoic Acid
Number analyzed (Participants) | 16 | 16
percentage of voice signal with tremor
  Baseline Magnitude of Acoustic Amplitude Tremor | 12.91 (6.46) | 13.49 (6.48)
  Post-test Magnitude of Acoustic Amplitude Tremor | 12.43 (7.37) | 9.35 (5.42)
  Baseline Magnitude of Acoustic Frequency Tremor | 5.57 (4.29) | 5.19 (3.58)
  Post-test Magnitude of Acoustic Frequency Tremor | 5.35 (3.76) | 3.98 (2.94)
Statistical Analysis 1: Comparison: Placebo vs Octanoic Acid; Separate measures for magnitude of amplitude tremor and magnitude of frequency tremor were analyzed as these variables can respond differently to treatment and may be differentially affected in essential voice tremor. Statistical modeling tested for post-treatment drug differences, with testing session as a repeated factor. Models were run with and without inclusion of baseline averages as a covariate per recommendations for cross-over treatment studies (Fleiss, Wallenstein & Rosenfeld, 1985); Test type: Superiority; p = 0.0216, Mixed Models Analysis — Statistical results for Magnitude of acoustic amplitude tremor. A priori significance threshold was set at P<0.05 for each of the two hypothesis-driven acoustic variables; This statistical test did not use the baseline scores as a covariate when comparing post-test scores between placebo and octanoic acid conditions
Statistical Analysis 2: Comparison: Placebo vs Octanoic Acid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0499, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; This statistical test used the baseline scores as a covariate when comparing post-test scores between placebo and octanoic acid conditions
Statistical Analysis 3: Comparison: Placebo vs Octanoic Acid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0339, Mixed Models Analysis — Statistical results for Magnitude of acoustic frequency tremor. A priori significance threshold was set at P<0.05 for each of the two hypothesis-driven acoustic variables; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Octanoic Acid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0450, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 3]; [statistical method as in outcome 1, analysis 2]

2. Secondary Outcome: Auditory-perceptual Tremor Severity Ratings
Description: Three experienced listeners independently rated each participant's voice from paired sample recordings comparing the baseline to post-test samples in randomized order for each condition. Sustained vowel and sentence-level recordings were rated, with decoded samples later analyzed for 1=better for post-test compared to baseline, 0= no difference between post-test and baseline. Maximum score for each participant was 3 (post-test was better for each of three raters). The range of possible scores was the sum of each of three raters' scores (0 to 3), with 0 indicating no difference between baseline and post-test voice tremor severity rating, and 3 indicating better voice (less tremor severity) at post-testing compared to pre-testing. Mean post-test values for task were compared for the octanoic acid and placebo conditions, and all raters were blind to which sample was a baseline versus a post-test recording, and which samples were associated with the [placebo or octanoic acid conditions.
Time Frame: Measured at baseline visits (1 & 2) and after 3 weeks of placebo or octanoic acid on post-test visits (1 & 2).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Octanoic Acid
Number analyzed (Participants) | 16 | 16
units on a scale
  Sustained vowel, summed binary ratings (0-3) | 1.25 (1.13) | 1.53 (1.13)
  Sentence-level, summed binary ratings (0-3) | 1.63 (1.12) | 1.19 (0.87)
Statistical Analysis 1: Comparison: Placebo vs Octanoic Acid; Statistical modeling tested for main effects of auditory-perceptual ratings for drug and task (sustained vowel and sentence-level ratings), and interaction effects of these variables. The summed scores, averaged across all participants, are provided separately for the sustained vowel and sentence-level ratings. Values range from 0 (no difference between baseline and post-test) to 3 (all three raters indicated that post-test sample was better (less tremor severity); Test type: Superiority; p = 0.7172, Mixed Models Analysis — A priori significance was set at P<0.05 for this hypothesis-driven auditory-perceptual variable. Main effect for drug is given above. For the main task effect, P=0.9602. For the interaction effect of drug*task, P=0.1699

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data were collected over approximately an 11 week period. This included data beginning with baseline testing in week 1, Phase 1 (placebo or octanoic acid condition) and continued through the week after post-test data was completed for Phase 2, on the final study visit (final nursing assessment visit).
Description: Participants completed symptom questionnaires with an independent nurse at four time-points: baseline before either the placebo or octanoic acid conditions, during the 3 weeks intake for each study phase, and upon completion of the study. Additionally, participants were called daily to inquire about any symptoms/symptom severity for three days after full drug intake was initiated for each study phase (placebo or octanoic acid) and then every 3-5 days thereafter each 3 week dosing period.
Groups:
- Placebo: Study phase 1 or 2, when participants were randomized to the 3-week intervention phase in which an inactive capsule (placebo or inactive drug) was taken once a day for 3 weeks.
- Octanoic Acid: Study phase 1 or 2, when participants were randomized to the 3-week intervention phase in which octanoic acid (the active drug) was taken once a day for 3 weeks.
Arm/Group | Placebo | Octanoic Acid
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 1/17 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Octanoic Acid (N=17)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No